CLINICAL TRIAL: NCT04198350
Title: Pancreatic Islet Transplantation to the Anterior Chamber of the Eye
Acronym: EYELETS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19SM5165
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes; Visual Impairment
Keywords: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Vision Disorders

STUDY DESIGN:
Intervention Model Description: This is a phase II prospective, interventional, open-labeled, proof-of-concept study.
  2 years per participant, 2 years 6 months in total Total n=6
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Islet implantation (Experimental)
  Interventions: Procedure: Islet implantation

INTERVENTIONS:
Procedure: Islet implantation — Transplantation of allogeneic pancreatic human islets will be performed into the anterior chamber of a single eye with the poorest visual acuity (see inclusion/exclusion criteria below). Up to 40 000 IEQ of islets in a maximum volume of 350µl will be transplanted.

SUMMARY:
This is a phase II prospective, interventional, open-labeled, proof-of-concept study.

2 years per participant, 2 years 6 months in total Total n=6

The primary objective is to assess the safety of human pancreatic islet transplantation into the ACE of participants with T1D.

Safety analyses will involve examination of the incidence, severity, and type of treatment emergent AEs reported, and changes in vital signs, ophthalmic status and laboratory test results from baseline (Day 0 pre-transplantation) to specified time points throughout the study.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is caused by the destruction of pancreatic islet cells through an autoimmune attack against insulin-producing beta cells in the endocrine pancreas. This in turn impairs glucose control causing multi-organ failure, morbidity and mortality which are also associated with high economic costs. While strict glucose control with insulin replacement therapy is the standard-of-care, achieving controlled glucose homeostasis remains a major challenge. Replacement of the insulin-producing beta cells through pancreatic islet transplantation has emerged as a promising therapy for T1D. Thus far, hundreds of islet transplantations have been performed in ongoing clinical trials worldwide. Islet transplantation is on the verge of obtaining FDA approval as a standard therapy in T1D. While ongoing clinical trials have focused on islet transplantation into the hepatic portal system, the search for alternative islet transplantation sites remains a priority for funding agencies and an active area of research. Studies have explored islet transplantation into different locations. One location of interest is the anterior chamber of the eye (ACE).

Importantly, these studies have shown several advantages offered by islet transplantation into the anterior chamber of the eye compared to other sites, which include:

* Local/topical immunosuppression and intervention potentially feasible.
* No IBMIR (Instant Blood Mediated Inflammatory Reaction) as when islets are injected to the portal vein with a major loss of islets.
* Good survival of transplanted islets due to limited anoxia time (fewer islets required to improve glycaemic control compared to other islet transplantation sites (i.e., liver)).
* Non-invasive monitoring/assessment of grafted islets with potential cellular resolution.
* Intraocular islets may function as "reporters" of native islets or islets transplanted elsewhere.
* Simpler surgical procedure as compared to other islet transplantation sites (i.e., liver).

Access to the ACE is a safe procedure routinely used by ophthalmic surgeons for the anterior segment surgery (e.g. cataract operations) and extraction of intraocular fluid for diagnostic purposes. Importantly, the ACE has unique immunological properties which regulate the immune system in such a way that allogeneic tissue placed in this compartment may be protected from immune rejection and this correlates with the generation of systemic immune tolerance through anterior chamber-associated immune deviation (ACAID) (Niederkorn and Streilein, 1982; Streilein and Niederkorn, 1985). Hence, the potential of inducing systemic immune tolerance and eliminating severe side-effects associated with systemic immunosuppression through local/topical drug application further highlight the significance and clinical relevance of this approach. Moreover, this introduces the possibility of transplanting additional islets elsewhere in the body without risk of rejection. Importantly, it was recently shown that islet grafts in the ACE also serve as "reporters" for the status of the pancreatic islets (Ilegems et al., 2013). This essentially demonstrates that islets in the ACE are reliable, easily accessible reporters for the overall health and islet function during interventions regimens aimed at regulating different aspects of the pancreatic islets.

INTERVENTION AND INDICATION

We intend to transplant six T1D participants with reduced vision in one or both eyes due to diabetes or other complications. Transplantation of allogeneic pancreatic human islets will be performed into the anterior chamber of a single eye with the poorest visual acuity (see inclusion/exclusion criteria below). Up to 40 000 IEQ of islets in a maximum volume of 350µl will be transplanted.

RATIONALE FOR THE INTENDED INTERVENTION

Improvement in glycaemic control is expected with the intended intervention, as measured with change in C-peptide, insulin, proinsulin and glucose levels during the MMTT, change in insulin requirements, change in HbA1c levels and in fasting glucose from baseline, change in total number of hypoglycaemic events, change of hypoglycaemia awareness, change in glycaemia fluctuations after transplant at Day 90, 180 and 365 post-operatively.

RISKS / BENEFITS

Successful islet transplantation reduces the risk to people with T1D of life-threatening hypoglycaemia and psychosocially debilitating glycaemic lability. While the long-term durability of these responses is at present uncertain, they persist for as long as some graft function is maintained, despite the eventual return to insulin therapy in the majority of islet transplant recipients in clinical trials of islet transplant in other sites. This partial function, as indicated by continued c-peptide production, may be present in as many as 80% of recipients after 5 years. Given our preliminary studies, however, a "marginal" islet mass in the anterior chamber of the eye may prove superior in conveying better function. Nonetheless, as long as graft function is maintained, fear of hypoglycaemia and anxiety are significantly lower after islet transplantation. Indeed, T1D participants with persistent c-peptide production have a significantly reduced risk of severe hypoglycaemia. Additionally, while most transplant recipients experience only a temporary reprieve from exogenous insulin therapy, a few have maintained insulin-independent graft function for more than 3 years. Shorter engraftment period in the anterior chamber of the eye may promote better survival of transplanted islets and lead to improved long-term graft function and further the duration of insulin-independence after transplantation, potentially leading to reductions in the secondary complications of T1D. At present, systemic immunosuppression is needed in all types of allogeneic organ- or cell transplantations. Due to the well-known side effects and risks involved with this medication the benefit from the procedure must out-weigh the risks. The benefit from the proposed treatment is unknown and therefore we have chosen participants that are already treated with immunosuppression not to lay this additional burden upon them.

Ophthalmic complications may include: elevated intraocular pressure, infection, corneal edema, severe inflammation, progression of diabetic retinopathy, or anterior segment neovascularization.

Only people with reduced VA in the treated eye and equal or better VA in the fellow eye will be included. Systemic complications due to the intervention are not expected. Nevertheless, systemic effects will be carefully monitored including possible immunization against the donor cells.

The proposed pilot study will mainly focus on the safety of islet transplantation to the ACE in a narrowly selected group of participants. However, if the study is successful we intend to treat participants with less severe disease and with broader systemic inclusion criteria. Ultimately, islet transplantation to the ACE may become an alternative route for cell therapy and disease monitoring in insulin-treated diabetes.

The islets will be transplanted into the eye with reduced vision to minimise any side-effects affecting your vision. The primary aim of the study is to evaulaute safety of the transplanting islets in the eye and regular eye examinations will be carried out throughout the study to identify any potential potential post-surgical risks caused by the transplanted islets which may include increased pressure in the eye, infection, swelling of the cornea, severe inflammation, progression of pre-existing diabetic retinopathy, or the formation of new blood vessels in the eye. To prevent these complications eye drops and antibiotics will be given. If needed a steroid injection can be administered to help with any issues and if necessary the transplanted islets will be removed.

JUSTIFICATION OF CHOICE OF STUDY POPULATION

Six people with T1D with reduced vision in one or both eyes due to diabetes or other complications, will be included in the study. Within this population we expect to identify participants with preserved anterior segment integrity which in turn reduces the risk of treatment-related complication. The choice of T1D participants facilitates evaluation of change in C-peptide and insulin levels. Islets may be surgically removed if uncontrolled complications cannot be managed non-surgically.

HYPOTHESIS

In this study, we aim to demonstrate safety and feasibility of pancreatic islet cell transplantation in the human eye. Also, its efficacy in restoring/improving glycaemic control should be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* T1D participants that fulfill criteria for islet transplantation
* Systemic immunosuppression
* At least one eye with VA from HM to 0.1, and fellow eye with equal or better VA
* Age ≥ 18 years
* Normal cornea with good visualization of the anterior segment
* Participant not eligible or with no wish for standard pancreatic islet into the hepatic portal system or pancreas transplantation
* Participants who have recently been involved in research or who are actively involved in research may be recruited at the discretion of the chief investigator if the active research has no impact on glucose self-management.

Exclusion Criteria:

* VA below HM or above 0.1
* Neovascular glaucoma
* Iris neovascularization
* Ongoing treatment with intraocular anti-VEGF or steroids (and no injection within 4 weeks) in the study eye and no anticipated need for therapy during study period.
* Ongoing retinal laser photocoagulation
* Signs of current infection or inflammation
* Intraocular surgery within 3 months
* Previous or planned anterior segment surgery for glaucoma
* Poor visualization of the anterior chamber

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Safety of the procedure with regards to opthalmic complications | 365 days
  Absence of ophthalmic complications (increased IOP, infection, severe inflammation in the treated or fellow eye, evidence of progression of diabetic retinopathy or anterior segment neovascularization) in the transplanted eye.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Oliver, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No